CLINICAL TRIAL: NCT02088463
Title: Efficacy of Lumbar Mobilization on Postpartum Low Back Pain in Egyptian Females: A Randomized Control Trial
Brief Title: Mobilization for Post Partum Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dr. Dalia Mohamed Kame, Associate Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/00368
Record Dates: First submitted 2014-03-05; First posted 2014-03-17 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain, Mechanical
Keywords: Mechanical LBP; Mobilization; Postpartum
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations; Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mobilization (manual therapy) (Experimental): Mobilization (manual therapy) posterior- anterior at the L3 for 2 minutes in addition to the traditional treatment in the form of infra-red and ultrasound. The treatment duration for the three groups was 3 times/week for 4 weeks.
  Interventions: Procedure: mobilization (manual therapy); Device: Ultrasound and infrared devices
- placebo mobilization (Placebo Comparator): placebo mobilization applied without force application. The treatment duration for the three groups was 3 times/week for 4 weeks
  Interventions: Procedure: Placebo mobilization; Device: Ultrasound and infrared devices
- Ultrasound and infrared therapy (Other): ultrasound and infrared are a traditional treatment for low back painThe treatment duration for the three groups was 3 times/week for 4 weeks.
  Interventions: Device: Ultrasound and infrared devices

INTERVENTIONS:
Procedure: mobilization (manual therapy) — mobilization is one of the manual therapy or treatments with the application of a gentle oscillatory passive movement to the spinal region specifically at the level of L3 in this study at the posterio-anterior direction.
  Other Names: PA mobilization
  Arms: Mobilization (manual therapy)
Procedure: Placebo mobilization — placebo mobilization is a tactile stimulation at the same level L3 without application of any force.
  Other Names: tactile stimulation
  Arms: placebo mobilization
Device: Ultrasound and infrared devices — ultrasound and infrared are the traditional treatment for low back pain , they are electrical modalities used in the field of physiotherapy to decrease the inflammation and the pain in musculoskeletal systems
  Other Names: US & IR

SUMMARY:
The study was conducted to the following purposes

1. To investigate the effect of lumbar mobilization on muscle activity in postpartum mechanical low back pain.
2. To investigate the effect of lumbar mobilization on pain intensity in postpartum mechanical low back pain patients.
3. To investigate the effect lumbar mobilization on functional disability in postpartum mechanical low back pain patients.
4. To compare between the effects of lumbar mobilization, tactile stimulation (placebo treatment) and traditional treatment in postpartum mechanical low back pain patients.

DETAILED DESCRIPTION:
all participants divided randomly into three groups, Group A (Study group) received PA lumbar mobilization plus traditional treatment which consisted of Ultrasonic and Infra-red. Group B (Placebo group) received placebo mobilization plus traditional treatment. Group C (Control group) received traditional treatment only

ELIGIBILITY:
Inclusion Criteria:

Females with LBP lasting more than 3 months since their delivery

* their age range 25-35 years old with body mass index (BMI) less than 30kg/m2

Exclusion Criteria:

* medical conditions that don't allow the subject to lie prone comfortably as, cardiovascular disease, uncontrolled hypertension, abdominal hernia, severe respiratory diseases, as well as problems in the back e.g. previous low back surgery, spinal malignancy. In addition to known rheumatic joint disease, and upper or lower motor neuron lesion that affects lower limbs

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-12; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | after 4 weeks from starting the intervention
  each case assessed two times pre- post intervention, intervention was lasted for 4 weeks
functional disability | after 4 weeks from starting the intervention
  each case assessed two times pre-post intervention, intervention lasted for 4 weeks
back muscle activity | after 4 weeks from starting the intervention
  each case assessed two time pre- post intervention, intervention lasted for 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dalia Shewitta, PhD, Principal Investigator — Assocciate Professor of Physical Therapy
Locations (1):
- Faculty of Physical Therapy, Cairo, Giza Governorate, Egypt